CLINICAL TRIAL: NCT02451501
Title: Influence of Body Posture on Pulmonary Aerosol Deposition
Acronym: NebuPostu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NebuPostu
Record Dates: First submitted 2015-05-07; First posted 2015-05-22 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Lying (Experimental): Nebulization in lying position
  Interventions: Device: AKITA
- Sitting (Active Comparator): Nebulization in sitting position
  Interventions: Device: AKITA

INTERVENTIONS:
Device: AKITA

SUMMARY:
To compare deposition in two different positions.

ELIGIBILITY:
Inclusion Criteria:

* Free of respiratory disease

Exclusion Criteria:

* Smokers

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Lung deposition by scintigraphy | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Reychler G, San Miguel-Pagola M, Aubriot AS, Herrero-Cortina B, Lecocq V, Hesse M, Liistro G, Jamar F. Targeted Lung Deposition From Nebulization Is Not Improved in the Lateral Decubitus Position in Healthy Volunteers. Respir Care. 2019 Dec;64(12):1537-1544. doi: 10.4187/respcare.06978. Epub 2019 Sep 10. PMID 31506338